CLINICAL TRIAL: NCT07084480
Title: Riesenzellarteriitis - Wege Zur "Precision Medicine"
Brief Title: Giant Cell Arteritis - Ways to Precision Medicine
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Riesenzellarteriitis-Register
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-07

CONDITIONS: Giant Cell Arteritis; Polymyalgia Rheumatic (PMR)
Keywords: non-interventional cohort study; aortic dilatation; innate lymhoid cells; optic coherence tomography; MRI
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Known patients: Patients, who are already known and had regular visits in the outpatient rheumatology department of the Würzburg university hospital. These patients already receive immunosuppressive therapy.
- New patients: Patients who have not yet been treated by the outpatient rheumatology department of the Würzburg university hospital, preferably but not limited to immunosuppressive therapy-naive patients.

SUMMARY:
Long-term follow-up of aortal adverse events, as well as glucocortioid-associated adverse events in patients with polymyalgia rheumatica (PMR) and giant cell arteritis (GCA).

DETAILED DESCRIPTION:
In this non-interventional cohort study the following aspects should be addressed:

* Can regular imaging procedures help to better assess the risk of aortic aneurysms and dissections over a period of 5-10 years after initial diagnosis of GCA?
* Which prognostic factors correlate with aortic events?
* What conclusions can be drawn about glucocorticoid-associated side effects over the longer (5-year) course?
* Can modern imaging in correlation with standardized clinical examination, serological markers and immunophenotypic testing define patient clusters within the clinically heterogeneous disease spectrum of GCA and PMR with the aim of individualizing therapy?
* What is the value of orbital MRI together with an ophthalmologic examination including fudoscopy and optical coherence tomography (OCT) in the detection of ischemic manifestations of GCA?
* Can a contrast agent-saving MRI technique (with 25 % less contrast agent) be used in GCA without impairing signal quality?
* Can rare lymphocyte populations be found by immunophenotyping, which provide information on the probability of recurrence or allow therapy control?

ELIGIBILITY:
Inclusion Criteria:

* Age greater or similar to 18 years
* Primary diagnosis of GCA or PMR

Exclusion Criteria:

* Age under 18 years
* lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GCA and PMR patients will be recruited in the department of rheumatology of the university hospital of Würzburg
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2033-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of aortic adverse events | Within 5 years
  Aortic adverse events include new foramation or progress of aortic aneurysms, and aortic dissection

SECONDARY OUTCOMES:
Incidence of glucocorticoid-related adverse events | within 5 years
  Assessment of the glucocorticoid toxicity index (GTI; excluding regular bone density measurements) to detect glucocorticoid-related adverse events.
  The GIT includes 1) a cumulative worsening score, which includes the cumulative glucocorticoid toxicity over time (minimum value of 0 and a maximum value of 439, a decrease is not possible) and 2) an aggregate improvement score, which allows for decreases and increases of toxicity (range from -346 to 439, with negative values indicating improvement and positive values indicating worsening of glucocorticoid toxicity)
Detection of ischemic complications in the eyes | within 5 years
  Is orbital MRI together with optic coherence tomography suitable to detect ischemic manifestations of GCA in the eye?
Performance of gadopiclenol in detecting vessel wall inflammation | within 5 years
  The contrast agent gadopiclenol should be evaluated for its use in MR angiography, i.e. if it depicts (peri) vessel wall inflammation equally to older contrast agents. In a sub-cohort of 20 % of the patients , MR angiographies will be performed with 25% reduced gadoplicenol.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gernert, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Universitätsklinikum Würzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No
single center study